CLINICAL TRIAL: NCT01159626
Title: A Phase 1, Randomized, Subject- and Investigator-blind, Sponsor-open, Placebo-controlled, Single- and Multiple-dose Escalation Study to Investigate the Pharmacokinetics, Safety and Tolerability of PF-03463275 in Healthy Male Japanese and Western Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability Study of PF-03463275 in Healthy Male Japanese and Western Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9131010
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Phase1; Pharmacokinetics; Healthy Male; Japanese; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 1-methyl-1H-imidazole-4-carboxylic acid (3-chloro-4-fluoro-benzyl)-(3-methyl-3-aza-bicyclo(3.1.0) hex-6-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (Experimental)
  Interventions: Drug: PF-03463275; Drug: Placebo
- Multiple dose (Experimental)
  Interventions: Drug: PF-03463275; Drug: Placebo

INTERVENTIONS:
Drug: PF-03463275 — Oral single 20 mg dose as two 10mg controlled release tablets
  Arms: Single dose
Drug: PF-03463275 — Oral single 40 mg dose as four 10mg controlled release tablets
  Arms: Single dose
Drug: PF-03463275 — Oral single 60 mg dose as six 10mg controlled release tablets
  Arms: Single dose
Drug: Placebo — Oral single dose as matching placebo
  Arms: Single dose
Drug: PF-03463275 — Oral multiple 40 mg doses as four 10mg controlled release tablets for 7 days
  Arms: Multiple dose
Drug: Placebo — Oral multiple doses as matching placebo for 7 days
  Arms: Multiple dose

SUMMARY:
This Phase 1 study is the first clinical trial in Japanese subjects. The study is designed to evaluate the single- and multiple-dose pharmacokinetics, safety and tolerability of PF-03463275 oral controlled release formulation in Japanese and Western male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2, and a total body weight >50 kg (110 lbs).
* Japanese subjects must have four Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Subjects that are genotyped to be PM (poor metabolizer), UM (ultrarapid metabolizer), IM/EM and EM/UM for CYP2D6 status.
* Evidence or history of clinically significant hematological (including anemia), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adverse events monitoring | Day 0 to Day 4 in each period of Cohort A, Day 0 to Day 10 in Cohort B
Vital signs, ECGs, clinical laboratory tests, clinical evaluations and examinations, suicidality assessment | Screening and Day 0 to Day 4 in each period of Cohort A, Screening and Day 0 to Day 10 in Cohort B
Serum (after single dose): Cmax, AUClast, AUCtau (Calculated only in Cohort B) and as data permit Tmax, AUCinf, t1/2 | Day 1 to Day 4 in each period of Cohort A, Day 1 in Cohort B
Serum (after multiple dose): Ctrough, Cmax*, AUCtau* and as data permit Tmax*, t1/2* and Rac* (accumulation ratio) * Calculated only after the last administration. | Day 2 to Day 10 in Cohort B

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9131010&StudyName=Pharmacokinetics%2C%20Safety%20and%20Tolerability%20Study%20of%20PF-03463275%20in%20Healthy%20Male%20Japanese%20and%20Western%20Subjects